CLINICAL TRIAL: NCT01410370
Title: Phase II Study of Continuous Endostar Infusion Combined With Radiotherapy for the Treatment of Patients With Brain Metastases
Brief Title: Continuous Endostar Infusion Combined With Radiotherapy in Patients With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Lianyungang (Other)
Responsible Party: Xiaodong Jiang, The First People's Hospital of Lianyungang
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Endu-201107
Record Dates: First submitted 2011-07-20; First posted 2011-08-05 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Brain Metastases
Keywords: Endostar; Radiotherapy; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Experimental): Radiotherapy plus Endostar
  Interventions: Radiation: 6MV-X ray; Drug: Endostar
- control (Active Comparator): Radiotherapy
  Interventions: Radiation: 6MV-X ray

INTERVENTIONS:
Radiation: 6MV-X ray — 3Gy/time, 5 times/week, a total of 10 times
Drug: Endostar — 7.5mg/m2/d, continuous infusion, in parallel with radiotherapy
  Arms: treatment

SUMMARY:
The aim of this study is to evaluate the clinical efficacy and safety of continuous Endostar infusion combined with radiotherapy for treatment of brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy with presence of intraparenchymal brain metastases
* Karnofsky performance status ≥ 40
* Measurable disease according to RECIST criteria
* Hematologic function: WBC ≥ 4.0×109/L, PLT ≥ 80×109/L, Hb ≥ 90g/L
* Renal function: Cr ≤ 2.0×ULN
* Hepatic function: BIL ≤ 2.0×ULN, ALT/AST ≤ 5.0×ULN
* Adequate cardiac function
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Evidence of bleeding diathesis or serious infection
* Serious cardiovascular disease (congestive heart failure, uncontrollable arrhythmia, unstable angina, myocardial infarction, serious heart valve disease, resistant hypertension)
* Uncontrollable mental and nervous disorders
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 month after initial treatment

SECONDARY OUTCOMES:
Overall Survival | 2 year
Serum VEGF Levels | at baseline and 1 month after initial treatment
VEGF levels in tumor tissue | at baseline and 1 month after initial treatment
Incidence of Adverse Events | up to 1 month after last dose
Cerebral Edema | 1 month after initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Jiang, MD, Principal Investigator — The First People's Hospital of Lianyungang
Locations (1):
- The First People's Hospital of Lianyungang, Lianyungang, Jiangsu, China